CLINICAL TRIAL: NCT05102240
Title: Developing Clinical High Efficiency Platforms for Individualised Treatment Through Integration of Advanced Radiation Technology, Quantitative Imaging and Molecular Biology and Machine Learning for Treatment of Cervix Cancer.
Brief Title: Development of Clinically High Efficient Platforms for Individualised Treatment of Cervix Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Tata Memorial Hospital (Other Government)
Collaborators: Bhabha Atomic Research Centre and Indian Institute of Technology, Mumbai. (Unknown); Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Supriya Sastri (chopra), Professor, Radiation Oncology, Tata Memorial Hospital
Other Study IDs: TMC IRB 900787; CTRI/2021/08/035810 (Registry Identifier: Clinical Trials Registry - India)
Record Dates: First submitted 2021-10-20; First posted 2021-11-01 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Cervix Cancer
Keywords: Advanced Radiation Technology; Quantitative Imaging; Molecular Biology; Machine Learning
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective study utilizing patient data to develop and validate Machine Learning application. Available imaging data sets of patients who have completed treatment will be used to develop Normal tissue complication probability and Tumour control probability

Hypothesis Integrating existing radiation treatment information, quantitative imaging and patient outcome data from completed and ongoing clinical trials will allow development of knowledge based systems for efficient treatment delivery and allow selection of patients for intensified treatment approaches in cervix cancer.

DETAILED DESCRIPTION:
For Aim 1. Automatic delineation of complex tumour targets for cervical cancer for the Gross Tumour Volume (GTV) at baseline and at brachytherapy and High Risk Clinical Target Volume(CTV) at baseline and brachytherapy will be done on MRI.

Following structures will be processed for automation on CT

1. Low Risk Clinical Target Volume (Low Risk CTV)
2. GTV: Nodal
3. Elective Nodal Pelvic Target Volume
4. Elective Nodal Pelvic and Paraaortic Volume
5. Rectum
6. Bladder
7. Sigmoid
8. Bowel
9. Bone Marrow

For Aim 2. The Investigator intend to employ machine learning for developing more robust normal tissue toxicity prediction models. Further advanced techniques like texture analysis of radiation dose maps and follow up tissue density will also be performed to develop predictive models of toxicity. By using our patient datasets, Investigator want to create a library of proton beam plans with the proton planning systems that will be available in department of radiation oncology and using the developed normal tissue complication plots available the information of achievable doses through protons can help in identifying patients who will benefit from proton therapy.

For Aim 3. Within this project Investigator intend to integrate staging, pathology and quantitative imaging texture features for response prediction and identification of "high risk cohort" in cervix cancer. Images and clinical data from patients that have MRI at baseline will be included The texture features can be used to categorise "good" and "poor responders" after chemoradiation. For the same cohort of patients the Investigator also have tissue available including results of additional biomarkers (like AKT,LICAM, PDL1,CD4 and CD8). The Investigator intend to first correlate difference in texture features and see if there is a pattern of different molecular features. In the second step imaging and molecular features could be integrated for developing" risk prediction models". GTV and HRCTV delineated on 150 data sets at baseline and brachytherapy within Aim 1 will be utilised to categorise responders and non-responders and validate another 150 patient data sets.

ELIGIBILITY:
Inclusion Criteria:

For Aim 1 and Aim 3:

* Patients treated within ongoing and completed clinical trials of chemoradiation and brachytherapy for cervix cancer with access to MRI/CT images at the time of diagnosis and brachytherapy For Aim 2
* Patients undergoing postoperative or definitive radiotherapy and treated within trials of postoperative or definitive RT.

Exclusion Criteria:

1. Lack of disease or toxicity outcomes.
2. Lack of images in the hospital database.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is about cervical cancer.
Study Population: Cervical cancer patients treated within ongoing and completed clinical trials of chemoradiation and brachytherapy for cervix cancer at our institute with access to MRI/CT images at time of diagnosis and brachytherapy, undergoing postoperative or definitive radiotherapy and treated within trials of postoperative or definitive RT.
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2022-02-24 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Generation of software for automated target delineation for cervix cancer | 3 years
  1. To develop and validate automated platforms for target delineation and planning for cervix cancer in time efficient manner through
  a. Machine learning based detection of abnormal cancerous tissues in multimodality medical diagnostic images.
  b . To train machine base systems for automated planning of external radiation and brachytherapy for gynaecological cancers.
Development and validation of Normal Tissue Complication Plots | 3 years
  2. To use existing databases and radiation dose maps, imaging texture features and adverse events data for machine learning to develop "normal tissue complication plots "and to identify cervix cancer patient subgroups that may benefit from advanced radiation techniques (like proton treatment)
Identify "high risk patient population" that may benefit from intensification of treatment in future | 3 years
  3. To use advanced image texture analysis within ongoing institutional and collaborative clinical trials to identify "high risk patient population" that may benefit from intensification of treatment in future

CONTACTS AND LOCATIONS:
Overall Officials: Supriya Sastri (nee Chopra), MD, Principal Investigator — Tata Memorial Centre, The Advanced Centre for Treatment, Research and Education in Cancer (ACTREC)
Locations (1):
- Advanced Centre of Treatment Research and Education In Cancer,Tata Memorial Centre, Navi Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Undecided